CLINICAL TRIAL: NCT06058975
Title: National Retrospective Study of Duodenal Trauma
Acronym: TRAUMADUOD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Urgences02
Record Dates: First submitted 2023-08-30; First posted 2023-09-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2023-09

CONDITIONS: Duodenal Diverticulization; Pyloric Exclusion; Gastrojejunostomy; Retrograde Duodenostomy; Distal Feeding Tube; Resection and Whipple Procedures; Primary Repairs
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Review the management of duodenal trauma in France

SUMMARY:
Duodenal injuries remain rare among abdominal trauma, concerning less than 5 % of cases. However, due to its central location, it is most commonly associated with multiple organs lesions, with the main three organs being the liver, the colon and the pancreas. Additionally, the penetrating mechanism is four times more common than blunt trauma and the most common duodenal site of injury is the second portion (36 %), the least being the first duodenum (13 %). These particularities generate a high morbidity, ranging from 22 to 27.1 %, and a mortality still as high as 5.3 to 30 % today. When facing it, surgeons are usually challenged in their strategy. Indeed, when surgery is required, different options can be chosen depending on the grade of the lesion and the involvement of the papilla and/or other organs. Primary repairs, duodenal diverticulization, pyloric exclusion, gastrojejunostomy, retrograde duodenostomy, distal feeding tube, or even resection and Whipple procedures, have all been described. Since the classification of the American Association for the surgery of trauma (AAST), most studies stratified their management as such: drainage only or primary repair for grade 1 and 2, jejunostomy and/or pyloric exclusion for grade 3, Whipple for grade 4 or 5. However, reviews of the literature aren't clear if this decisional tree is in correlation with lower morbidities, and often different procedures have been reported for the same grade. The escalation of technical exclusions among severe grades became controversial. As an example, pyloric exclusion has been criticized in its preventive role of protecting the suture, being useless at least, or even worse at times. Thus, in the recent years, the management has been focused towards minimization. Indeed, in the retrospective review of the Pan-American trauma society primary repair alone was performed in 80 % of cases, all grades comprised. Although mortality was high, duodenal suture line leak was statistically lower among survivors over every grade.

To clear the situation, prospective studies are difficult if not impossible in such context. Thus, The investigators propose this national benchmark, to retrospectively review in France the management of duodenal trauma, depending on the grade, and its associated morbidity.

ELIGIBILITY:
Inclusion Criteria:

* patients with duodenal trauma,
* older than 18 years old.

Exclusion Criteria:

* pregnancy
* previous duodenal surgery.
* Associated surrounding organs trauma, was not an exclusion criterion, but duodenal trauma must have been one of the main injuries.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with duodenal trauma
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 1 month after trauma
  Study mortality is overall mortality, not specific to abdominal trauma. It corresponds to grade 5 of the Clavien-Dindo classification.
Specific mortality | 1 month after trauma
  Specific mortality is the mortality due to abdominal trauma, including abdominal compartment syndrome, coagulopathy, hemorrhage, multi-organ failure, etc. It excludes brain death, mortality due to trauma of other body regions. It corresponds to grade 5 of the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Severe morbidity | 3 months after trauma
  Morbidity will be recorded according to the Clavien-Dindo classification. We will study overall morbidity and severe morbidity (stages 3 and 4). As a reminder, stage 1 corresponds to a simple deviation from the operative course, stage 2 to medical treatment, stage 3 to interventional management (with or without general anaesthesia), and stage 4 to organ or multi-visceral failure.
Kind of treatment: medical, endoscopic or surgical | The first 3 months after trauma
  We will record the type of initial treatment performed, whether non-operative, endoscopic, laparoscopic or by laparotomy.
  We will collect the results of this initial treatment, including the possibility of complementary treatments, whatever the approach used and any failures.
  Non-operative management is defined as an exclusive medical attitude, including diagnostic imaging, but without interventional procedures.
  Interventional radiology management is defined as a percutaneous procedure performed under the control of diagnostic imaging, e.g. ultrasound- or scan-guided puncture of a collection.
  Endoscopic management includes diagnostic or therapeutic endoscopy, for example: endoscopic realignment of the Wirsung duct, puncture of a pancreatic pseudocyst, duodenal stenting, etc.
  Surgical management is defined as any surgical procedure requiring an opening of the abdomen. The approach is indicated as laparotomy or laparoscopy.
type of injury of the duodenum | no later than the 7th day after the trauma
  The surgeon is free to describe the lesions, in order to gather as much information as possible on the location of the lesion, its size, etc.
  We will also ask investigators to describe the lesions encountered, using the classification established by the AAST (American Association for the Surgery of Trauma).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frey S, Bentellis I, Gaujoux S, Girard E, Abba J, Chirica M, Bertrand M, Boutry E, Mege D, Aubert M, Alves A, Hornez E, Mulliri A, Brustia R, Hentati H, Lauka L, Laurent A, Sommacale D, Turco C, Dezeustre M, Bajul M, Castel A, Facy O, Grellet R, Sulpice L, Menegaux F, Delestre M, Lermite E, Monchal T, Amrou R, Bacoeur-Ouzillou O, Pezet D, Bonnet J, Buc E, Passot G, Schneck AS, Birnbaum DJ, Blanc PY, Le Roy B, Monneuse O, Rodriguez Q, Suc B, Baque P, Dubuisson V, Massalou D. How are duodenal trauma managed? A French nationwide study. World J Emerg Surg. 2025 Dec 9;20(1):89. doi: 10.1186/s13017-025-00661-z. PMID 41366408